CLINICAL TRIAL: NCT06583876
Title: Bio Refine for Functional Mitral Regurgitation - a Safety & Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bio Refine Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-6470
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-09

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Coriofix treatment (Experimental)
  Interventions: Device: Coriofix System

INTERVENTIONS:
Device: Coriofix System — Treatment of functional mitral regurgitation by reducing the mitral valve annular area through ablation of the posterior annulus.

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Bio Refine Coriofix System and determine if it might help in treatment of functional mitral regurgitation.

The study will include patients with symptomatic secondary mitral regurgitation in whom mitral surgery cannot and/or will not be offered as a treatment option (the risk is prohibitive).

Potential patients will be screened to confirm that all inclusion/exclusion criteria are met, with final eligibility confirmation on day of procedure.

All enrolled subjects who went through the procedure will be followed during the procedure to hospital discharge.

Additional follow up time points are scheduled at 30 days, 6 months and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Local heart team has determined that mitral valve surgery will not be offered as a treatment option
* Symptomatic secondary mitral regurgitation (3+ or 4+)
* Adequately treated in compliance with optimal guideline-directed medical therapy for heart failure for at least 90 days
* NYHA functional class II, III or ambulatory IV
* LVEF ≥30%.
* Written informed consent has been obtained

Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization.
* CABG, PCI or TAVR within the prior 90 days.
* Aortic or tricuspid valve disease requiring surgery or transcatheter intervention or severe tricuspid regurgitation.
* COPD requiring continuous home oxygen therapy or chronic outpatient oral steroid use.
* CVA or TIA within prior 180 days.
* Hypotension
* Any history of ventricular arrythmia
* Patients implanted with any kind of CIED
* Life expectancy <12 months due to non-cardiac conditions
* Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
* TEE is contraindicated or high risk
* Pregnant or planning pregnancy within next 12 months
* Currently participating in an investigational drug or another device study that has not reached its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Coriofix System Safety | 30 days
  Absence of Major Device- or Procedure-Related Serious Adverse Events

SECONDARY OUTCOMES:
Coriofix System Safety | 6 and 12 months
  Absence of Major Device- or Procedure-Related Serious Adverse Events
Device technical success | Procedure
  Successful system operation with no related emergency surgery or reintervention
Treatment success | 30 days
  Change of MR grade

CONTACTS AND LOCATIONS:
Locations (4):
- Gottsegen National Cardiovascular Center, Budapest, Hungary
- Rabin Medical Center, Petah Tikva, Israel
- Serbia (2):
  - Institute for Cardiovascular Diseases "Dedinje", Belgrade
  - University Clinical Center Kragujevac, Kragujevac

IPD SHARING:
Plan to Share IPD: No